CLINICAL TRIAL: NCT04759768
Title: Two-Period, Two-Treatment, Randomized Crossover Study of the Pharmacokinetics of Nalmefene by Intranasal and Intramuscular Administration in Healthy Volunteers
Brief Title: Pharmacokinetic Evaluation of Intranasal Nalmefene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opiant Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPNT003-PK-001
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Nalmefene (Experimental): Nalmefene hydrochloride nasal spray, 3mg, 1 spray
  Interventions: Drug: Nalmefene Hydrochloride
- Intramuscular Nalmefene (Active Comparator): Nalmefene injection, 1mg, 1 injection
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene Hydrochloride — 3mg nasal spray
  Arms: Intranasal Nalmefene
Drug: Nalmefene — 1mg intramuscular injection
  Arms: Intramuscular Nalmefene

SUMMARY:
This study is to determine the pharmacokinetics (how the body absorbs, breaks down and eliminates drug from your body) of nalmefene when given intranasally (IN;into the nose) compared to a dose of nalmefene when given intramuscularly (IM; into the muscle); to compare the blood levels of nalmefene when given IN to nalmefene when given IM; and to evaluate the safety and tolerability of nalmefene IN.

DETAILED DESCRIPTION:
Open-label, randomized, 2-period, 2-treatment, 2-sequence, crossover study in 68 healthy volunteers. Subjects will be assigned to each of the 2 possible sequences. Each subject will receive 2 treatments during the 2 dosing periods: Intranasal (IN) dose of 3 mg nalmefene hydrochloride and intramuscular (IM) dose of 1.0 mg nalmefene, with a 4 day washout period between doses. Screening can occur up to 28 days before baseline admission, subjects will then stay in the inpatient facility for 7 days to complete the treatment phase of the study and will be discharged following completion of the discharge procedures at the end of the last period. Subjects will be called 3 to 5 days after discharge to inquire concerning Adverse Events (AEs) and concomitant medications since discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years inclusive
* BMI ranging from 18 to 30 kg/m2, inclusive
* Adequate venous access
* Subjects must be non-smokers

Exclusion Criteria:

* History of clinically significant disease
* Significant trauma injury, major surgery, open biopsy within 30 days prior to screening
* Following an abnormal diet 4 weeks prior to screening
* Use of over the counter medications, dietary supplements, herbal products, vitamins or opioid analgesics 14 days before intervention
* Use of enzyme altering drugs 30 days before intervention
* Use of nasal products 28 days before intervention and throughout the study
* Previous or current opioid, alcohol, or other drug dependence
* Donated or received blood 30 days before intervention
* Women who are pregnant or breastfeeding at screening
* Women of childbearing potential unless surgically sterile or use effective contraception
* Current or recent upper respiratory tract infection
* Allergic to nalmefene

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bass, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crystal R, Ellison M, Purdon C, Skolnick P. Pharmacokinetic Properties of an FDA-approved Intranasal Nalmefene Formulation for the Treatment of Opioid Overdose. Clin Pharmacol Drug Dev. 2024 Jan;13(1):58-69. doi: 10.1002/cpdd.1312. Epub 2023 Jul 27. PMID 37496452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Complete
Groups:
- Intranasal Nalmefene Then Intramuscular Nalmefene: 3 mg nalmefene hydrochloride intranasally (1 spray) then 1 mg nalmefene hydrochloride solution intramuscularly (single dose)
- Intramuscular Nalmefene Then Intranasal Nalmefene: 1 mg nalmefene hydrochloride solution intramuscularly (single dose) then 3 mg nalmefene hydrochloride intranasally (1 spray)
Period: First Intervention (1 Day)
Arm/Group | Intranasal Nalmefene Then Intramuscular Nalmefene | Intramuscular Nalmefene Then Intranasal Nalmefene
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Intranasal Nalmefene Then Intramuscular Nalmefene | Intramuscular Nalmefene Then Intranasal Nalmefene
Started | 34 | 34
Completed | 34 | 32
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Second Intervention (1 Day)
Arm/Group | Intranasal Nalmefene Then Intramuscular Nalmefene | Intramuscular Nalmefene Then Intranasal Nalmefene
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Nalmefene Then Intramuscular Nalmefene | Intramuscular Nalmefene Then Intranasal Nalmefene | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Customized [Count of Participants; unit: Participants]
  Age 18 to 55 years old | 34 | 34 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 24 | 16 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Black or African American | 11 | 12 | 23
  Native Hawaiian or other specific islander | 1 | 0 | 1
  White | 21 | 20 | 41
  Multiple | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.58 (2.540) | 25.60 (2.996) | 26.09 (2.800)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum concentration of plasma nalmefene comparing IN to IM
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intranasal Nalmefene | Intramuscular Nalmefene
Number analyzed (Participants) | 66 | 68
ng/ml | 12.2 (6.71) | 1.77 (1.18)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum concentration of plasma nalmefene comparing IN to IM
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Intranasal Nalmefene | Intramuscular Nalmefene
Number analyzed (Participants) | 66 | 68
hours | 0.25 [0.0833 to 2] | 0.333 [0.117 to 18]

3. Primary Outcome: Area Under the Curve (AUC-inf)
Description: Area under the curve of plasma nalmefene comparing IN to IM
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Groups:
- Intranasal Nalmefene: 3 mg nalmefene hydrochloride intranasally (1 spray)
- Intramuscular Nalmefene: 1 mg nalmefene hydrochloride solution intramuscularly (single dose)
Arm/Group | Intranasal Nalmefene | Intramuscular Nalmefene
Number analyzed (Participants) | 66 | 68
hour*ng/mL | 41.5 (8.45) | 17.0 (3.13)

4. Primary Outcome: Half-life (t1/2)
Description: Half life of plasma nalmefene comparing IN to IM
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Intranasal Nalmefene | Intramuscular Nalmefene
Number analyzed (Participants) | 66 | 68
hour | 11.4 (2.37) | 10.6 (1.95)

ADVERSE EVENTS:
Time Frame: Subjects in the study from baseline to 7 days with a =3 to 5 day follow-up
Arm/Group | Intranasal Nalmefene | Intramuscular Nalmefene
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 42/66 | 8/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Nalmefene (N=66) | Intramuscular Nalmefene (N=68)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 37 | 0
headache (Nervous system disorders) | 3 | 4
nausea (Gastrointestinal disorders) | 2 | 4
dizziness (Nervous system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04759768/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04759768/SAP_001.pdf